CLINICAL TRIAL: NCT06104826
Title: Health-related Quality of Life Outcomes and Bleeding Rates Among Patients With Severe Hemophilia A on Emicizumab: Real World Data
Brief Title: Health-Related Quality of Life Outcomes and Bleeding Rates Among Patients With Severe Hemophilia A on Emicizumab
Acronym: ML43518
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Newark Beth Israel Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Narang Shalu, Associate Clinical Professor, Rutgers New Jersey and Robert Wood Johnson Medical School, Newark Beth Israel Medical Center
Other Study IDs: 2023.20
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Hemophilia A
Keywords: Bleeding Disorder; Hemophilia; Quality of Life Outcomes; Emicizumab
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders | interventions — emicizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Emicizumab — Emicizumab in Hemophilia A

SUMMARY:
The main purposes of this study are to determine if use of emicizumab prophylaxis treatment reduces number of bleeding episodes, if it improves quality of life of individuals and if improves arthropathy in persons with hemophilia A.

DETAILED DESCRIPTION:
The main purpose of this study is to determine if use of emicizumab prophylaxis treatment reduces number of bleeding episodes and if it affects quality of life of individuals with hemophilia.

Patients with hemophilia A, especially those with severe disease, have recurrent bleeding in joints, muscles and deep tissue and recurrent bleeding in the same joint can result in irreversible damage in bone and cartilage and lead to disabling arthropathy. Treatment involves replacement with exogenous recombinant factor concentrates that can prevent further bleeding episodes but not the ongoing joint damage. In addition, treatment with recombinant factor concentrates can lead to inhibitory antibodies resulting in inability to use those for further treatment. The burden of this disease on patients and caregivers is well recognized.

Participant will be asked about bleeding episodes needing additional factor replacement in addition to checking bleeding log prior to starting emicizumab and at additional times after starting emicizumab. In addition, investigators would ask participant to complete questionnaire about participant's and/or their caregiver's quality of life prior to starting emicizumab and at additional times after starting emicizumab. Participant will also have joint scores measured before and at additional times after starting emicizumab. All the information collected will remain confidential and would only be shared with members of study team.

ELIGIBILITY:
Inclusion Criteria Part A: ABR

* Signed Informed Consent/Assent Form
* Age 4 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Diagnosis of hemophilia A (any severity) on emicizumab or factor concentrate prophylaxis for at least 12 months each
* Plan to be adherent to emicizumab prophylaxis during the study
* Patient with inhibitors
* Patient without inhibitors Part B: HRQoL and Arthropathy
* Signed Informed Consent/Assent Form
* Age 4 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Diagnosis of hemophilia A (any severity) who has decided to switch to emicizumab prophylaxis
* Plan to be adherent to emicizumab prophylaxis during the study
* Individuals of childbearing age will be included in this study. Their participation involves voluntary completion of a questionnaire. There are no additional precautions required for this population.
* Patient/parent must be able to read and write English/Spanish

Exclusion Criteria:

* Part A: ABR

  * Patients who are on a clinical trial for prophylaxis
  * Patients with other bleeding disorders needing any scheduled treatment
  * No eligibility restrictions will be based on gender, race, ethnic background or economic status

Part B: HRQoL and Arthropathy

* Patients who are on a clinical trial for prophylaxis
* Patients with other bleeding disorders needing any scheduled treatment
* Patients/parents who refuse to complete questionnaire or have joint health assessment by HJHS
* No eligibility restrictions will be based on gender, race, ethnic background or economic status

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include children and adults who are males and females with hemophilia A for all parts of the study. Children and adults are equally at risk for bleeding and hence we would collect information about bleeding events in both children and adults on emicizumab or on factor concentrates to calculate ABR. There will be no exclusion based on race or ethnicity. For HRQoL part of the study, children and their families will be included.The Quality of life was found to be poor both among children affected with hemophilia and their parents and perceived impact on family. Hemophilic arthropathy can be seen in children and adults and therefore, this outcome must be studied in both populations as it can be disabling at any age.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To obtain and compare the annual bleeding rate in patients with hemophilia A on emicizumab before and after being on emicizumab. | 12 months
  Annualized Bleeding Rates (ABR)
To evaluate the health related quality of life in patients with hemophilia A before and after being on emicizumab. | 12 months
  Quality of Life Questionaries
To study any clinical changes in arthropathy. | 12 months
  Joint score measurements

SECONDARY OUTCOMES:
To study practitioner's preference for emicizumab schedule and how it affects compliance | 12 months
  ABR

CONTACTS AND LOCATIONS:
Locations (1):
- Newark Beth Israel Medical Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided